CLINICAL TRIAL: NCT05529342
Title: A Long-Term Follow-Up Study of Participants Treated With the Lentiviral-Based Genetically Modified, Autologous Cell Product, AGT103-T
Brief Title: Long-term Follow-up of Study Participant Treated With Lentiviral-Based Genetically Modified Autologous Cell Product ,AGT103-T
Status: Enrolling by invitation | Type: Observational
Sponsor: American Gene Technologies International Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AGT103-T-LTFU
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: HIV
Keywords: Long term follow-up; Genetically modified CD4 T cells; Gene Therapy; Lentivirus vector

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Gene modified therapy — No investigational cell product will be administered

SUMMARY:
Long-term follow-up of study subjects who received AGT103-T product in HIV study. The AGT103-T is genetically modified cells that resist infection with HIV causing a depletion of HIV in HIV-infected study participants.

DETAILED DESCRIPTION:
The primary objective of this study is to monitor study participant who receive the genetically modified gag specific CD4 T cells for the long term adverse event, evaluate sustained impact on immunity and the persistence of vector modified CD4 T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Received the investigational product, AGT103-T, in the AGT-sponsored AGT-HC168 clinical trial
2. Provided written informed consent, signed and dated by the study participant in the long-term follow-up study

Exclusion Criteria:

1. Did not receive the investigational product, AGT103-T

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject who received the investigational product AGT103-T in the AGT-HC168 clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2038-05-23 (Estimated); Study Completion 2038-09-29 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence of delayed adverse events (AE) to gene therapy | 1year to 15years post infusion
  The presence of malignancies, incidence or exacerbation of pre-existing neurologic disorder, new incidence or exacerbation of a prior rheumatologic or other autoimmune disorder, the new incidence of a hematologic disorder post infusion with AGT103T

SECONDARY OUTCOMES:
The persistence and the immunity impact of the vector-modified T cells | 1year to 15 years
  Evaluate sustained impact on immunity measured by CD4 T cell responses to Gag peptides Measure proportion of participants with absence of replication competent lentivirus (RCL) Measure persistence of vector-modified cells (transgene copies per CD4 T cell)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Georgetown University, Washington D.C., District of Columbia
  - Washington Health Institute, Washington D.C., District of Columbia